CLINICAL TRIAL: NCT01730391
Title: Neisseria Meningitidis Burden of Disease
Brief Title: Neisseria Meningitidis Burden of Disease Study
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 114989
Record Dates: First submitted 2012-11-15; First posted 2012-11-21 (Estimated); Last update posted 2015-11-11 (Estimated); Status verified 2015-11

CONDITIONS: Streptococcus Pneumoniae; Neisseria Meningitidis; Haemophilus Influenzae
MeSH Terms: conditions — Haemophilus Infections | interventions — Data Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Cerebrospinal Fluid (CSF) sample (collected as part of routine practice)

GROUPS / COHORTS (1):
- Study cohort: Subjects visiting the hospital with suspected bacterial meningitis in The Philippines and Vietnam.
  Interventions: Other: Data collection; Other: CSF samples testing

INTERVENTIONS:
Other: Data collection — Collection of demographic data and vaccination history
Other: CSF samples testing — CSF samples will be tested for the determination of N. meningitidis and other likely bacterial pathogens that cause bacterial meningitis (S. pneumoniae and H. influenzae)

SUMMARY:
This study aims to provide an estimate of the proportion of suspected cases of bacterial meningitis that are due to N. meningitidis and the serogroup responsible in The Philippines and Vietnam.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes can and will comply with the requirements of the protocol or subjects who the investigator believes that parent(s)/Legally Acceptable Representative(s) [LAR(s)] can and will comply with the requirements of the protocol.
* Written informed consent obtained from the subject/from the parent(s)/LAR of the subject.
* A male or female subject who visits the hospital with suspected bacterial meningitis.
* CSF sample taken as part of routine practice.

Exclusion Criteria:

* Child in care.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects visiting the hospital with suspected bacterial meningitis in The Philippines and Vietnam.
Sampling Method: Non-Probability Sample
Enrollment: 521 (Actual)
Dates: Start 2013-01; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Prevalence of N. meningitis in CSF samples | At enrollment (Day 0)
Serogroup of N. meningitis positive samples | At enrollment (Day 0)

SECONDARY OUTCOMES:
Further characterization of N. meningitidis using Multi Locus Sequence Typing | At enrollment (Day 0)
Prevalence of Haemophilus influenzae and Streptococcus pneumoniae in CSF samples as causes of bacterial meningitis | At enrollment (Day 0)
Serotype of Streptococcus pneumoniae positive samples | At enrollment (Day 0)
Further classification of Haemophilus influenzae positive samples into Type B and non-B Types | At enrollment (Day 0)
Total number of subjects with suspected bacterial meningitis (according to diagnostic criteria used by each participating hospital to identify this condition) | At enrollment (Day 0)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- Philippines (2):
  - GSK Investigational Site, Baguio City, Benguet
  - GSK Investigational Site, Quezon City
- GSK Investigational Site, Hanoi, Vietnam